CLINICAL TRIAL: NCT06676618
Title: Effect of Multimodal Exercise Training on Disease Activity and Functional Status in Patients With Multiple Sclerosis
Brief Title: Effect of Multimodal Exercise Training in Patients With Multiple Sclerosis
Acronym: PwMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Pelin Vural, Lecturer, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IU-C20204-161
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Physiotherapy; Degenerative diseases; Disease activity; Multimodal
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Exercise Training Group (Experimental): Participants in the multimodal exercise training group will be given a treatment protocol consisting of aerobic exercise and strengthening exercises in the presence of a physiotherapist for a total of 12 weeks, 3 days a week for 1 hour.
  Interventions: Other: Multimodal Exercise Training
- Control Group (Other): Participants in the control group will be put on the waiting list after all assessment methods have been applied and will be re-evaluated at the end of 12 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Multimodal Exercise Training — The exercise training consisting of aerobic, strengthening and balance exercises will be applied for 12 weeks/3days for 1hour. One day of the exercise training will be performed in a clinical environment with a physiotherapist, and the other 2 days of the week, participants will be asked to apply asynchronous video-based telerehabilitation over the internet in their own homes. The asynchronous video-based telerehabilitation application will be performed through an account created specifically for the participant on the "www.telenororehab.com" website. The exercise program will be created according to the individual's condition and progression will be provided every 3 weeks. Patients who do not attend 3 consecutive sessions will be excluded from the study.
  Arms: Multimodal Exercise Training Group
Other: Control Group — Participants in the control group will be placed on the waiting list after all evaluation methods have been applied and will be re-evaluated at the end of 12 weeks. After the evaluations, individuals in the control group will also be given multimodal exercise training.
  Arms: Control Group

SUMMARY:
The study aims to examine the effects of multimodal exercise training including aerobic, strengthening and balance exercises via face-to-face and asynchronous video-based telerehabilitation on disease activity, disability level, aerobic capacity, physical activity level, balance, fatigue level and quality of life in individuals with multiple sclerosis. Therefore, this study consists of two hypotheses.

Hypotheses:

H0: Multimodal exercise training has no effect on disease activity and functional status in patients with multiple sclerosis H1: Multimodal exercise training has effects on disease activity and functional status in patients with multiple sclerosis

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a leading cause of disability in young adults, with symptoms varying based on lesion size, location, and disease course. These symptoms often worsen over time, significantly impacting quality of life. To manage symptoms and potentially affect disease activity, patients are often directed to exercise interventions, though the impact on disease progression is still being studied. Neuroimaging, particularly magnetic resonance imaging (MRI), is commonly used to monitor MS, but MRI does not reveal brain activation levels, which is why functional MRI is recommended for a more detailed evaluation. Exercise, both face-to-face and telerehabilitation (TR), is considered an effective treatment for MS. Studies show that TR increases patient adherence and can be as effective as in-person therapy. Our study aims to assess the effects of a multimodal exercise program combining face-to-face and TR on disease activity and functional status in patients with MS (PwMS). PwMS with an Expanded Disability Status Scale (EDSS) score of 3.0 to 5.5 will be randomly assigned to either the multimodal exercise training group (Group I) or a control group (Group II). Disease activity, disability, aerobic capacity, physical activity, balance, fatigue, and quality of life will be evaluated. Group I will participate in exercise training three days a week (one day in-person, two days TR) for 12 weeks. Group II will receive no exercise during this period and will be reassessed after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with multiple sclerosis by a neurologist
* Volunteering to participate in the study
* Being ambulatory
* EDSS between 3.0-5.5
* Being literate
* Having internet access
* Not having participated in a standardized physiotherapy and rehabilitation program in the last 3 months

Exclusion Criteria:

* Having an orthopedic problem affecting its mobility
* Having psychiatric problems, severe cognitive impairment, or epilepsy in addition to the MS diagnosis
* Blurred vision or visual impairment
* Pregnancy
* Having had an attack or received corticosteroid treatment 3 months before participating in the study
* Having a disease affecting immunological parameters (infection, cancer, etc.)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Functional Composite Test (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  The Multiple Sclerosis Functional Composite Test evaluates disease activity through three sections: cognitive status, and upper and lower extremity function. The Paced Auditory Serial Addition Test (PASAT) measures auditory processing speed, attention, flexibility, and calculation by having the patient add numbers presented at three-second intervals. The score is based on correct answers, with a maximum of 60 points. The Timed 25 Foot Walking Test (T25FWT) assesses lower extremity function by recording the time (in seconds) taken to walk 7.62 meters as quickly and safely as possible, with the average of two trials used for scoring. The 9-Hole Peg Test (9DPT) evaluates upper extremity function by having the patient place and remove nine pegs as quickly as possible, with scores based on the average of two trials for each hand.
Functional Magnetic Resonance Imaging (fMRI) (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  fMRI is a non-invasive method that allows the examination of central nervous system function and the identification of abnormal activation patterns and/or functional connectivity caused by diseases (Rocca et al 2024).In our study, functional MRI evaluations are planned to be performed using parallel imaging sequences with a 3 T Siemens device with a 32-channel head coil. High-resolution (1 x 1 x 1 mm isotropic) sagittal 190 slices will be obtained with a T1-weighted imaging sequence (TR/TE: 7.7/3.7 ms;, FA: 8°; FOV: 256 x 256). Functional resting state data will be taken with a single-shot echo planar imaging (EPI) sequence consisting of 35 slices of 4 mm thickness, 300 dynamic shots (TR/TE: 2230/30 ms, FA: 77°; matrix: 80x80) and will last approximately 11 minutes. Before functional acquisition, magnetic field maps will be recorded in order to correct signal distortions caused by tissue inhomogeneities in the magnetic field during the analysis phase.
Brain-derived neurotrophic factor (BDNF) assessment (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  BDNF is a neurotrophin that affects the survival, growth and function of neurons in the central and peripheral nervous system, provides stabilization of synapses, and regulates synaptic function, axon and dendrite branching. In our study, Enzyme-Linked Immunosorbent Assay (ELISA) will be used to assess the BDNF levels of participants. All participants will be asked not to consume alcohol and caffeine in the last 12 hours before blood collection, not to take any anti-inflammatory drugs other than their routine treatments and not to exercise. The blood samples to be collected will be centrifuged and stored at -80 degrees in Eppendorf or Falcon tubes (15 ml) (Shobeiri et al 2022; Briken et al. 2016). After the treatments are completed, the blood taken will be analyzed by experienced technicians in the laboratory together with the blood taken before exercise training.

SECONDARY OUTCOMES:
The Expanded Disability Status Scale (EDSS) (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  EDSS will be used to assess the disability level of the participants. The scale widely used to assess the level of disability in PwMS, evaluates 8 functional subsystems. These systems consist of pyramidal functions, cerebellar functions, brainstem functions, sensory functions, bladder-bowel functions, visual functions, cognitive functions, and other functions. The scale consists of a 20-category ordinal rating system ranging from 0 (normal neurological examination regardless of symptoms) to 10 (death due to MS), with 0.5-point increments starting from 1 (Kurtzke 1983).
6 Minute Walk Test (6MWT) (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  It is a simple, practical test applied according to the standard protocol of the American Thoracic Society (ATS) to measure walking capacity. It has been reported that the test is valid and reliable in MS patients with mild and moderate disability. In our study, 6MWT will be performed in accordance with the standards set in the guidelines for MS patients. The participant will be asked to walk as fast as possible at his own walking pace on the 30-meter track for 6 minutes. Before starting the test, participants will be explained that they can rest if they develop excessive fatigue or respiratory distress during the test and that this time is included in the test period. As a result of the test, the distance traveled by the participant will be recorded in meters (Paltamaa et al. 2005; ATS statement 2002).
ActiGraph wGT3X-BT (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  Accelerometer is a valid, reliable and objective measurement device that measures the number, intensity and energy consumption of activities. The device can be attached to the wrist and ankle with an elastic belt. In our study, the amount of physical activity and energy consumption of the participants in a week will be assessed using ActiGraph wGT3X-BT Accelerometer (Polhemus et al. 2022).
The Godin Leisure-Time Exercise Questionnaire (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  It is a self-reported questionnaire with two questions that measures the physical activity behavior of the participants. In the first question, the frequencies of mild, moderate and intense physical activity performed for more than 15 minutes in a normal week are questioned. Weekly frequencies of light, moderate, and vigorous physical activities are multiplied by 3, 5 and 9 metabolic equivalents, respectively, and the sum of the results is recorded as total leisure activity. Second question seeks the frequency of activity that causes sweating in a normal week is questioned. Less than 14 scores means insufficiently active/sedentary, 14-23 scores means moderately active and 24 scores or more means active. So higher scores better outcomes (Weikert et al. 2010).
Balance Assessment (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  Our study will evaluate static and dynamic balance. The One-Legged Standing Test is a reliable test that can be easily applied to evaluate static balance. For this test, the participant will be asked to stand on the right and left feet respectively. As a result of the test, the time the participant can stand on one leg will be recorded in seconds (Fry & Pfalzer 2006). The Timed Up and Go Test is a test used to evaluate dynamic balance. The test measures the time it takes for a person to get up from a chair, walk 3 meters at a comfortable pace, return to the chair and sit down in seconds. The test starts when the participant gets up from the chair and ends when he/she sits back down on the chair. A shorter time represents better mobility (Cattaneo et al. 2006).
Fatigue Severity Scale (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  It is a scale that evaluates the fatigue of MS patients in daily functions. In the evaluation made with 9 questions, each question is scored between 1 (totally disagree) - 7 (totally agree). The result score is the average value of nine questions. High score indicates increased severity of fatigue (Krupp et al. 1989).
Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) (The change between the initial value and the value after 3 months will be evaluated). | Baseline and end of weeks 12
  The scale consists of 31 questions in 6 subgroups including physical condition, symptoms, psychological condition, self, relationship with friends, family and medical personnel. The answers are scored between 0 and 5 and a score ranging from 0 to 100 is obtained. Higher scores indicate higher quality of life (Simeoni et al. 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Vural, MSc, Principal Investigator — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Yonca Zenginler Yazgan, PhD, Study Chair — Istanbul University-Cerrahpasa Faculty of Health Science; Murat Kürtüncü, Prof. Dr., Study Chair — Istanbul University Istanbul Faculty of Medicine Department of Neurology
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)

REFERENCES:
- [Background] Rocca MA, Romano F, Tedone N, Filippi M. Advanced neuroimaging techniques to explore the effects of motor and cognitive rehabilitation in multiple sclerosis. J Neurol. 2024 Jul;271(7):3806-3848. doi: 10.1007/s00415-024-12395-0. Epub 2024 May 1. PMID 38691168
- [Background] Shobeiri P, Karimi A, Momtazmanesh S, Teixeira AL, Teunissen CE, van Wegen EEH, Hirsch MA, Yekaninejad MS, Rezaei N. Exercise-induced increase in blood-based brain-derived neurotrophic factor (BDNF) in people with multiple sclerosis: A systematic review and meta-analysis of exercise intervention trials. PLoS One. 2022 Mar 3;17(3):e0264557. doi: 10.1371/journal.pone.0264557. eCollection 2022. PMID 35239684
- [Background] Briken S, Rosenkranz SC, Keminer O, Patra S, Ketels G, Heesen C, Hellweg R, Pless O, Schulz KH, Gold SM. Effects of exercise on Irisin, BDNF and IL-6 serum levels in patients with progressive multiple sclerosis. J Neuroimmunol. 2016 Oct 15;299:53-58. doi: 10.1016/j.jneuroim.2016.08.007. Epub 2016 Aug 5. PMID 27725121
- [Background] Cutter GR, Baier ML, Rudick RA, Cookfair DL, Fischer JS, Petkau J, Syndulko K, Weinshenker BG, Antel JP, Confavreux C, Ellison GW, Lublin F, Miller AE, Rao SM, Reingold S, Thompson A, Willoughby E. Development of a multiple sclerosis functional composite as a clinical trial outcome measure. Brain. 1999 May;122 ( Pt 5):871-82. doi: 10.1093/brain/122.5.871. PMID 10355672
- [Background] Bosma LV, Kragt JJ, Brieva L, Khaleeli Z, Montalban X, Polman CH, Thompson AJ, Tintore M, Uitdehaag BM. Progression on the Multiple Sclerosis Functional Composite in multiple sclerosis: what is the optimal cut-off for the three components? Mult Scler. 2010 Jul;16(7):862-7. doi: 10.1177/1352458510370464. Epub 2010 May 20. PMID 20488826
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Polhemus A, Haag C, Sieber C, Sylvester R, Kool J, Gonzenbach R, von Wyl V. Methodological heterogeneity biases physical activity metrics derived from the Actigraph GT3X in multiple sclerosis: A rapid review and comparative study. Front Rehabil Sci. 2022 Nov 28;3:989658. doi: 10.3389/fresc.2022.989658. eCollection 2022. PMID 36518351
- [Background] Weikert M, Motl RW, Suh Y, McAuley E, Wynn D. Accelerometry in persons with multiple sclerosis: measurement of physical activity or walking mobility? J Neurol Sci. 2010 Mar 15;290(1-2):6-11. doi: 10.1016/j.jns.2009.12.021. Epub 2010 Jan 8. PMID 20060544
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Simeoni M, Auquier P, Fernandez O, Flachenecker P, Stecchi S, Constantinescu C, Idiman E, Boyko A, Beiske A, Vollmer T, Triantafyllou N, O'Connor P, Barak Y, Biermann L, Cristiano E, Atweh S, Patrick D, Robitail S, Ammoury N, Beresniak A, Pelletier J; MusiQol study group. Validation of the Multiple Sclerosis International Quality of Life questionnaire. Mult Scler. 2008 Mar;14(2):219-30. doi: 10.1177/1352458507080733. Epub 2007 Oct 17. PMID 17942521